CLINICAL TRIAL: NCT01343693
Title: A Post Market Surveillance Validation to Evaluate the Effectiveness of the MaxAn Anterior Cervical Plate
Brief Title: MaxAn Post Market Surveillance Validation
Acronym: MaxAn
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-059
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: DDD; Deformity; Tumor; Fracture
Keywords: DDD; Deformity; Tumor; Fracture; Cervical
MeSH Terms: conditions — Congenital Abnormalities; Neoplasms; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anterior cervical discectomy and fusion: Any subject with DDD, tumor, deformity ot trauma to the cervical spine in which the investigator determines the subject will require an ACDF using the MaxAn Plate.

SUMMARY:
This study is being performed to document the outcomes of subjects using our MaxAn Anterior Cervical Plate and assess them for Adjacent level Disease. All subjects will be followed for 2 years.

DETAILED DESCRIPTION:
The purpose of this Post Market Surveillance Validation is to document the performance and clinical outcomes of the MaxAn® Anterior Cervical Plate System. Dr. Park, et.al conducted a retrospective review and found a positive association between adjacent-level ossification following anterior cervical plate procedures and the plate-to-disc distance. 1 They concluded that when the anterior cervical plates were placed at least 5mm away from the adjacent disc spaces, there was a decrease in the likelihood of moderate-to-severe adjacent-level ossification. The design of the MaxAn Anterior Cervical Plate and accompanying technique allows this type of plate placement; therefore we will be looking at the radiographic outcomes of these subjects and comparing them to the retrospective chart review conducted by Dr. Park using the MaxAn Technique allows you to achieve plate placement of 5mm from the supraadjacent level which will help minimize the risk of adjacent level ossification.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo a one to three-level primary spinal fusion surgery between the levels of C2-T1 (Cervical 2 to Thoracic 1) using the MaxAn® Anterior Cervical Plate System.
* Subject has agreed to participate in this study, sign the informed consent and have agreed to return for the 6, 12 and 24 month follow-up visits.
* Subjects or their representative must be willing and able to give informed consent.

Exclusion Criteria:

* Subject has spinal infection or inflammation at any level.
* Subject is morbidly obese, defined as a BMI greater than 40.
* Subject has a mental illness, alcoholism or drug abuse.
* Subject has a metal sensitivity/foreign body sensitivity.
* Subject has inadequate tissue coverage over the operative site.
* Subject has an open wound local to the operative area, or rapid joint disease, bone absorption, osteopenia and/or osteoporosis.
* Female subjects who are pregnant or plan to become pregnant in the next 24 months or who are lactating.
* Subject who does not meet the specific indications for use of the MaxAn® Anterior Cervical Plate System.
* Subjects participating in another clinical research study.
* Any previous cervical spinal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This post market surveillance study will enroll two hundred (200) subjects across 10 clinical centers within the United States with subjects followed for 24 months post-surgery. All subjects enrolled in the study will be recruited from the pool of subjects presenting to each investigational site for an anterior cervical fusion procedure. The 10 surgeons chosen to participate in this study will be thoroughly knowledgeable in the medical, surgical and mechanical aspects of the MaxAn® Anterior Cervical Plate System. The following inclusion and exclusion criteria must be met for a patient to be considered eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2011-06; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Dix, MD, Principal Investigator — Maryland Spine and Brain
Locations (6):
- United States (6):
  - Montgomery Spine Center, Montgomery, Alabama
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Community Neurosurgery, Indianapolis, Indiana
  - Maryland Spine and Brain, Annapolis, Maryland
  - Cary Orthopedics, Cary, North Carolina
  - DFW Center for Spinal Disorders, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ACDF With MaxAn Plate: Any subject with DDD, tumor, deformity ot trauma to the cervical spine in which the investigator determines the subject will require an ACDF using the MaxAn Plate.
Period: Overall Study
Arm/Group | ACDF With MaxAn Plate
Started | 119
Completed | 110
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | ACDF With MaxAn Plate
Number analyzed (Participants) | 119
Age, Continuous [Mean (Full Range); unit: years] | 54.3 [31.4 to 81.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 119
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (5.5)
Employment Status [Count of Participants; unit: Participants]
  Currently Working | 50
  Disabled/Retired Due to Ill Health | 28
  Retired | 23
  Unemployed | 7
  Workers Compensation | 3
  Not Reported | 8
Tobacco Use [Count of Participants; unit: Participants]
  Current | 37
  Past | 30
  Never | 52
Previous Cervical Spine Surgery [Count of Participants; unit: Participants] — History of any previous spine surgery in the cervical region, included fusion, discectomy, decompression, laminectomy.
  Participants
    Yes | 24
    No | 95
Number of Operated Levels [Count of Participants; unit: Participants]
  One vertebral level | 27
  Two vertebral levels | 69
  Three vertebral levels | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Differing Severity of Adjacent Level Ossification
Description: Qualitatively assessed by an independent Radiologist using lateral radiographs Grade 0 - None Grade 1 - Mild (if the ossification extended across <50% of the disc space) Grade 2 - Moderate (if the ossification extended across ≥ 50% of the disc space) Grade 3 - Severe (if there is complete bridging of the adjacent disc space)
Time Frame: 24 Months
Population: Ten of the 110 patients with 24 month follow up were not evaluated for this endpoint. Eight had missing radiographs and 2 had unevaluable radiographs.
Measure: Count of Participants; unit: Participants
Arm/Group | ACDF With MaxAn Plate
Number analyzed (Participants) | 110
Participants
  Grade 0 | 36
  Grade 1 | 38
  Grade 2 | 16
  Grade 3 | 10
  Unable to Assess | 2
  Missing Radiographs | 8

2. Secondary Outcome: Change in Neck Disability Index (NDI)
Description: The Neck Disability Index (NDI) is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain', with the points summed to a total score. The test can be interpretated as a raw score, with a minimum score of 0 and a maximum score of 50. A higher score indicates more patient-rated disability. To use the NDI for patient decisions, a clinically important change was calculated as 5 points.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACDF With MaxAn Plate
Number analyzed (Participants) | 110
score on a scale | 22.0 (20.0)

ADVERSE EVENTS:
Time Frame: 24 Months
Description: All adverse events, including both observed or volunteered problems, complaints, symptoms, physical signs or disease which either occur during the study, having been absent at baseline, or, if present at baseline, appear to worsen during the clinical outcomes collection study were recorded as part of the study.
Arm/Group | ACDF With MaxAn Plate
All-Cause Mortality (participants affected / at risk) | 0/119
Serious Adverse Events (participants affected / at risk) | 14/119
Other Adverse Events (participants affected / at risk) | 83/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACDF With MaxAn Plate (N=119)
Neck pain (Musculoskeletal and connective tissue disorders) | 14 (16) — Subsequent surgery due to neck pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACDF With MaxAn Plate (N=119)
Musculoskeletal Other - Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 20 (20)
Musculoskeletal other - Degenerative disc disease (Musculoskeletal and connective tissue disorders) | 15 (15)
Neck Pain (Musculoskeletal and connective tissue disorders) | 14 (14)
Paresthesia (Nervous system disorders) | 8 (8) — Upper extremity numbness
Radiculitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) — Cervical radiculopathy
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) — Shoulder pain
Dysphagia (Gastrointestinal disorders) | 9 (9)
Headache (Nervous system disorders) | 6 (6)
Wound complication (Injury, poisoning and procedural complications) | 4 (4)
Procedural complication, other (Injury, poisoning and procedural complications) | 2 (2) — Subsidence of spine implant
Procedural complication other (Injury, poisoning and procedural complications) | 1 (1) — Migration of spine implant
Radiculitis (Musculoskeletal and connective tissue disorders) | 7 (7) — Lumbar radiculopathy
Musculoskeletal other (Musculoskeletal and connective tissue disorders) | 3 (3) — Lumbar spondylosis
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT01343693/Prot_SAP_000.pdf